CLINICAL TRIAL: NCT07319065
Title: Left Ventricular Myocardial Work for Predicting Response to Cardiac Resynchronization Therapy (CRT): A Multi-Center Study
Brief Title: Left Ventricular Myocardial Work for Predicting Response to CRT
Acronym: CARE-MW
Status: Not yet recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: CARE-MW Study; General Electric Healthcare (Other Grant/Funding Number: General Electric Healthcare Systems Trade Development (Shanghai) Co., Ltd.)
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: CRT Non-Response; LBBB; HF - Heart Failure; Healthy Adult
Keywords: Myocardial work
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Adults Group: Healthy adults aged 18 to 79 years are planned to be stratified into 6 age groups: 18-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years, and ≥70 years. Each age group will include 120 participants of each sex.
- Patients with heart failure and left bundle branch block who are scheduled to undergo CRT treatment: Ultrasound machine LVEF ≤ 35%; QRS ≥ 150ms; LBBB; Optimal drug therapy for at least 3 months before implantation 600 participants
  Interventions: Diagnostic Test: Ultrasound machine
- Patients with LBBB who have preserved LVEF: LVEF≥53%； LBBB 600 participants
  Interventions: Diagnostic Test: Ultrasound machine
- Patients with reduced LVEF but without LBBB: LVEF ≤ 35%, non-LBBB 600 participants
  Interventions: Diagnostic Test: Ultrasound machine

INTERVENTIONS:
Diagnostic Test: Ultrasound machine — Myocardial work is a recently developed non-invasive method that incorporates the LV afterload into the overall longitudinal strain (GLS) analysis of echocardiography. Myocardial work reflects the contractile ability of the heart, stroke work per beat, residual myocardial contractile ability, myocardial oxygen consumption, useless work, and useful work, which is represented by the pressure-volume loop analysis and thus has the potential to predict the efficacy of CRT.
  Groups: Patients with LBBB who have preserved LVEF; Patients with heart failure and left bundle branch block who are scheduled to undergo CRT treatment; Patients with reduced LVEF but without LBBB

SUMMARY:
This study aims to establish the normal reference values for left ventricular myocardial work in healthy Chinese adults and the influencing factors. Non-invasive myocardial work serves as a new parameter for identifying CRT responders and provides a scoring system for predicting the efficacy of CRT in clinical practice. CRT can improve cardiac function and quality of life, and reduce mortality and hospitalization rates due to heart failure (HF). Currently, the number of CRT treatments is increasing year by year, but even when strictly following the indications, approximately 30% of patients do not respond. Therefore, precise prediction of CRT efficacy is of great clinical significance for improving prognosis. Currently, the indications for CRT mainly rely on clinical, electrocardiogram (CLBBB), and LVEF. By correcting ventricular contraction asynchrony to improve systolic function, however, CLBBB indicates electrical asynchrony, and LVEF improvement depends on mechanical synchrony. If the mechanical asynchrony of the ventricles can be evaluated directly before surgery, it will help predict the efficacy of CRT. Myocardial work is a recently developed non-invasive method that combines LV afterload with the overall longitudinal strain (GLS) analysis of echocardiography. Myocardial work reflects the contraction ability of the heart, stroke work, residual myocardial contraction ability, myocardial oxygen consumption, useless work, useful work, etc., and is represented by the pressure-volume loop analysis, thus having the potential to predict the efficacy of CRT. Therefore, this study intends to adopt the left ventricular myocardial work technique, combined with the current indication criteria, to predict the long-term efficacy of patients with heart failure who are scheduled for CRT treatment, thereby increasing the response rate of CRT and improving the prognosis of patients. Currently, there are no normal reference values for left ventricular myocardial work in healthy Chinese adults. Therefore, our center has initiated this multicenter clinical research project, collaborating with multiple ultrasound centers across the country, aiming to establish the normal ultrasound values for left ventricular myocardial work in healthy Chinese adults, providing new quantitative reference basis for the diagnosis of myocardial function, assessment of the severity of myocardial lesions, and efficacy observation.

ELIGIBILITY:
Healthy Adults Group

Inclusion Criteria:

* Participants must meet all of the following criteria to be enrolled:

  1. Of Han Chinese ethnicity
  2. Aged 18-79 years
  3. Normal blood pressure (< 140/90 mmHg)
  4. Normal fasting blood glucose
  5. Normal blood lipid levels (triglycerides, total cholesterol, low-density lipoprotein, high-density lipoprotein)
  6. Normal complete blood count results (hemoglobin concentration, white blood cell count, red blood cell count, platelet count)
  7. Normal liver and renal function (alanine transaminase < 2× upper limit of normal; normal creatinine and blood urea nitrogen)
  8. Normal electrocardiogram results (occasional atrial premature beats may be enrolled at the investigator's discretion)
  9. No structural heart disease and normal cardiac function confirmed by echocardiography

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

1. Clinically significant cardiac valve regurgitation (≥ mild severity)
2. Respiratory diseases: acute or chronic respiratory disorders
3. Endocrine diseases: thyroid disease, diabetes mellitus, hyperaldosteronism, pheochromocytoma, etc.
4. Abnormal liver function (alanine transaminase > 2× upper limit of normal), abnormal renal function (elevated creatinine beyond normal range), or dyslipidemia (elevated triglycerides, total cholesterol, low-density lipoprotein, or high-density lipoprotein)
5. Other systemic diseases: anemia, malignancy, connective tissue disease, large artery/peripheral vascular diseases (aortic dilation, aortic dissection, coarctation of the aorta, Takayasu arteritis, atherosclerosis), etc.
6. Pregnant or lactating women
7. Professional athletes
8. Poor-quality ultrasound images that cannot support parameter measurement and analysis

Heart failure patients with LBBB who are scheduled for CRT treatment Group

Inclusion criteria:

1. LVEF ≤ 35%
2. QRS ≥ 150ms; LBBB
3. At least 3 months of optimal drug therapy before implantation

Exclusion Criteria:

1. Suffering from connective tissue diseases such as systemic lupus erythematosus, polymyositis, and rheumatoid arthritis;
2. Having a history of blood diseases and severe systemic diseases such as infections;
3. Those who cannot cooperate with the examinations.

Patients with LBBB who have preserved LVEF Group

Inclusion criteria:

1. LVEF≥53%
2. LBBB

Exclusion Criteria:

1. Suffering from connective tissue diseases such as systemic lupus erythematosus, polymyositis, and rheumatoid arthritis;
2. Having a history of blood diseases and severe systemic diseases such as infections;
3. Those who cannot cooperate with the examinations.

Patients with reduced LVEF but without LBBB Group

Inclusion criteria:

1. LVEF ≤ 35%
2. non-LBBB

Exclusion Criteria:

1. Suffering from connective tissue diseases such as systemic lupus erythematosus, polymyositis, and rheumatoid arthritis;
2. Having a history of blood diseases and severe systemic diseases such as infections;
3. Those who cannot cooperate with the examinations.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolls 4 groups (18-79 years) from clinics/community:
  Healthy Adults: Han Chinese with normal cardiovascular function (vitals, labs, ECG, echo; no structural heart disease/systemic diseases/poor ultrasound).
  Heart failure patients with LBBB who are scheduled for CRT treatment： LVEF ≤ 35%,QRS ≥ 150ms; LBBB.At least 3 months of optimal drug therapy before implantation.
  Patients with LBBB who have preserved LVEF :LVEF≥53%, LBBB. Patients with reduced LVEF but without LBBB :LVEF ≤ 35%,non-LBBB.
Sampling Method: Probability Sample
Enrollment: 3240 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall work index（GWI） | At study enrollment (baseline)
  The curve area representing the left ventricular PSL from the closure of the mitral valve to its opening, that is, the overall contractile work of the myocardium

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, MD, Principal Investigator — First Hospital of China Medical University
Locations (82):
- China (82):
  - Anhui University of Chinese Medicine First Affiliated Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wannan, Anhui
  - The Provincial Hospital Affiliated to Fuzhou University, Fuzhou, Fujian
  - Fujian Provincial Geriatric Hospital, Guizhou, Fujian
  - Guizhou Provincial People's Hospital, Guizhou, Fujian
  - Union Hospital Affiliated to Fujian Medical University, Guizhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The First Hospital of Qinhuangdao City, Qinhuangdao, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Longnan Hospital of Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Heinan
  - FuWai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan Medical University (Xinxiang Medical University), Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Enshi Central Hospital, Enshi, Hubei
  - Puai Hospital of Wuhan City / The Fourth Hospital of Wuhan City, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Hospital of Traditional Chinese Medicine, Hubei Province, Xiangyang, Hubei
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - The First People's Hospital of Lianyungang City, Lianyungang, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First People's Hospital of Nantong City, Nantong, Jiangsu
  - The Third People's Hospital of Nantong City, Nantong, Jiangsu
  - Suqian Hospital of Jiangsu Provincial People's Hospital, Suqian, Jiangsu
  - The Hospital of Traditional Chinese Medicine of Suzhou City, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The People's Hospital of Wuxi City, Wuxi, Jiangsu
  - Su Bei People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Guizhou Medical University, Guizhoucun, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Jilin, Jilin
  - The Second Hospital of Jilin University, Jilin, Jilin
  - Central Hospital of Anshan City, Anshan, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Golden Autumn Hospital, Shenyang, Liaoning
  - Shengjing Hospital, China Medical University, Shenyang, Liaoning
  - Chifeng Hospital, Chifeng, Neimenggu
  - The People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Jinan Central Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Bethea Hospital of Shanxi Province, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital (Shanxi Cardiovascular Hospital Research Institute), Taiyuan, Shanxi
  - The Cancer Hospital of Shanxi Province, Taiyuan, Shanxi
  - The People's Hospital of Shanxi Province, Taiyuan, Shanxi
  - Tangdu Hospital, Air Force Medical University, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Xindu District People's Hospital of Chengdu City, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - The People's Hospital of Ya'an City, Ya'an, Sichuan
  - Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine / The Fourth Affiliated Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - Dianxi Central Hospital of Yunnan Province, Dingxi, Yunnan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lihuili Hospital of Ningbo Medical Center, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The Second Hospital of Ningbo City, Ningbo, Zhejiang
  - The Second Hospital of Shaoxing City, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The People's Hospital of Zhuji City, Zhuji, Zhejiang
  - The First Hospital of Peking University, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Shanghai Chest Hospital, Shanghai
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang

IPD SHARING:
Plan to Share IPD: No